CLINICAL TRIAL: NCT02272348
Title: Evaluation of Self-management of Patients With Type 1 Diabetes After Education to Functional Insulin Therapy
Brief Title: Self-management of Type 1 Diabetes Under Functional Insulin Therapy
Acronym: EVAUTODIAB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in methodology too important - end of randomization
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9372
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes; Basal-bolus Multiple-dily Insulin Injections; Insulin Pump (CSII)
Keywords: Therapeutic education; Functional insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education to functional insulin therapy immediately (Experimental): Immediately after inclusion, patients will follow a functional insulin therapy training course during 2.5 days.
  Interventions: Other: Training course to functional insulin therapy
- No education to functional insulin therapy immediately (Other): After inclusion in the study, patients go on usual diabetes management. At the end of study, they will receive education to functional insulin therapy.
  Interventions: Other: Usual diabetes management.

INTERVENTIONS:
Other: Training course to functional insulin therapy — Carbohydrate counting, carbohydrate/insulin ratio, sensitivity to insulin factor
  Arms: Education to functional insulin therapy immediately
Other: Usual diabetes management.
  Arms: No education to functional insulin therapy immediately

SUMMARY:
Therapeutic education of patients is a mandatory component of intensive insulin therapy of type 1 diabetes in order to reach optimal safety and efficacy. Used educational methods aim at facilitating patients' autonomy in their own management of diabetes. Therefore, self-management of patient with type 1 diabetes must be systematically assessed in order to evaluate the effectiveness of education programs .The main objective of this prospective controlled randomized monocentric study is to assess the impact of functional insulin therapy on the level of self-management of patients with type 1 diabetes via Confidence In Diabetes Self-care scale (CIDS) test.

DETAILED DESCRIPTION:
170 patients with type 1 diabetes, volunteering for education to functional insulin therapy, will be recruited by the Department od Endocrinology, Diabetes, Nutrition of Montpellier University Hospital.

After inclusion, the patients will be randomized in 2 groups: group 1 will be immediately trained to functional insulin therapy and group 2 will be trained at the end of the study. The patients will be met as outpatients 3 months after inclusion. The primary endpoint will be the global score for CIDS questionnaire.

Secondary endpoints will include: HbA1c level at month 3, frequency of hypoglycemia from inclusion to month 3, scores for each of the 20 items of CIDS questionnaire.

An ancillary study will assess: the acceptability of the new EAD questionnaire which specifically evaluates the self-management of diabetes, the concordance validity of EAD and CDIS questionnaires, the reproducibility test-retest, the internal consistency and the sensitivity to change of EAD questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes from at least 1 year
* Age from 18 to 70 (70 not included)
* Basal-bolus multiple-dily insulin injections or insulin pump (CSII)
* Informed consent
* Affiliated or benefit from an insurance regimen

Exclusion Criteria:

* Type 2 diabetes
* Unable to make mathematic calculation
* Pregnancy, breast-feeding or absence of effective contraception
* Psychiatric and/or cognitive status uncompatible with study
* Eating disorders
* Law protected person, vulnerable person

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
To assess the impact of therapeutic education by functional insulin therapy in patients with type 1 diabetes on their ability to disease self-management. | three months (from inclusion until end of study)
  CIDS questionnaire

SECONDARY OUTCOMES:
To assess the effect of education to functional insulin therapy on HbA1c level | three months (from inclusion until end of study)
  HbA1c
To assess the effect of education to functional insulin therapy on hypoglycemia frequency | three months (from inclusion until end of study)
  Hypoglycemia occurrence
To assess the effect of education to functional insulinotherapy on the score of each of the 20 items of CIDS questioonaire | three months (from inclusion until end of study)
  CIDS questionnaire sub scores
To assess the validity, the concordance and the sensitivity to change of EAD questionnaire (specific for self-management of diabetes) in comparison with CIDS test | three months (from inclusion until end of study)
  EAD questionnaire score

CONTACTS AND LOCATIONS:
Overall Officials: Elise DUTERTRE, MD, Principal Investigator — CHU Montpellier, France
Locations (1):
- Lapeyronie Hospital - CHU de Montpellier, Montpellier, France